CLINICAL TRIAL: NCT03664206
Title: Assessing Motor Neuron Disease Pathophysiology by Two Novel Methods - Threshold Tracking Transcranial Magnetic Stimulation and Magnetic Resonance Spectroscopy
Brief Title: Assessing Motor Neuron Disease Mechanisms by Threshold Tracking Transcranial Magnetic Stimulation and Magnetic Resonance Spectroscopy
Status: Withdrawn | Type: Observational
Why Stopped: The part on MRS could not be completed
Sponsor: Sándor Beniczky (Other)
Collaborators: Lundbeck Foundation (Other); Aage og Johanne Louis-Hansens Fond (Other); The A.P Moeller Foundation for Advancement of Medical Science (Unknown); Danish Council for Independent Research (Other); Aarhus University Hospital (Other); Central Denmark Region (Other)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: AMND; 7025-00066B (Other Grant/Funding Number: Independent Research Fund Denmark); 18-2B-2454 (Other Grant/Funding Number: Aage og Johanne Louis-Hansens Fond); 17-L-0365 (Other Grant/Funding Number: The A.P. Møller Foundation); 3530 (Other Grant/Funding Number: Lundbeck Foundation)
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Cortical Excitability
Keywords: Treshold Tracking Transcranial Magnetic Stimulation; Magnetic Resonance Spectroscopy; Inter-rater agreement; Reproducibililty of Results; Case-control Studies; Biomarkers; Intra-rater agreement
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: MRS, conventional TMS and treshold tracking TMS
  The participants will be told not to consume coffee or alcohol or do exhausting exercise 12, 24 and 48 hours, respectively, prior to the examinations
  Interventions: Diagnostic Test: MRS, conventional TMS and treshold tracking TMS
- Healthy subjects: MRS, conventional TMS and treshold tracking TMS
  The participants will be told not to consume coffee or alcohol or do exhausting exercise 12, 24 and 48 hours, respectively, prior to the examinations
  Interventions: Diagnostic Test: MRS, conventional TMS and treshold tracking TMS

INTERVENTIONS:
Diagnostic Test: MRS, conventional TMS and treshold tracking TMS — Using
  * two MagStim 200 magnetic stimulator and a figure-of-eightc double 70 mm coil
  * SPECIAL MR Spectroscopy sequence
  In addition, each group will undergo neurological examination

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a motor neuron disease, which cases the death of neurons controlling the voluntary muscles. The death of motor neurons leads eventually to muscle weakness and muscle atrophy and as a consequence thereof, ALS patients die in average within three years after symptom onset due to respiratory failure.

No cure for ALS is currently known, and the medical diagnosis and clinical treatment are impeded by the lack of reliable diagnostic tools for objective disease assessment, and by the limited insight in disease pathophysiology since the underlying disease mechanisms still have not been fully elucidated.

An unbalance in the concentrations of GABA and glutamate, the most important inhibitory and excitatory brain metabolites, is suggested to play a role in the disease mechanisms of ALS. By applying Magnetic Resonance Spectroscopy (MRS), a magnetic resonance method which allows for quantification of brain metabolites, GABA and glutamate concentration can be quantified and thus hopefully elucidate their role in ALS disease mechanism.

Threshold Tracking Transcranial Magnetic Stimulation (TT-TMS) studies carried out by a single research group have demonstrated cortical hyperexcitability (a physiology state in which neurons in the cerebral cortex are easier activated) as an early feature in ALS patients. For this reason, TT-TMS was suggested as a biomarker of ALS by the research group. However, to be able to suggest a test as a biomarker, one must show the test is reliable and reproducible.

The objectives of this study are therefore: to explore the pathophysiology of ALS by investigating the interaction between neuronal networks as assessed by TT-TMS and conventional TMS and MRS, and to investigate the reliability and reproducibility of TT-TMS. The aim is to examine the utility of TT-TMS and MRS as diagnostic tools for objective detection of ALS in the early disease stage.

The study will include 60 participants in total, subdivided into two groups: 30 healthy participants and 30 patients with clinical suspicion of motor neuron disease or ALS. Each participant will undergo examination with TMS and MRS, the primary outcomes will be compared between the two groups and the results from the TMS examinations and the MRS-scans will be correlated.

ELIGIBILITY:
Inclusion Criteria:

Patients with

* possible, probable or definite ALS according to international criteria;
* progressive muscular atrophy;
* clinical suspicion of motor neuron disease or ALS

Healthy participants: no younger than 45 years of age

Exclusion Criteria:

Patients and healthy participants:

* ealier central or peripheral nervous system disease
* pacemaker or other implants
* pregnancy
* use of medications known to affect central nervous system

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited among patients examined at the Department of Neurophysiology who are referred for diagnostic neurophysiological examinations without any relation to the proposed project and at the Department of Neurology who are being examining for routine controls.
  The healthy participants will be recruited by announcement at the homepage www.forsoegsperson.dk/ and by announcement at Aarhus University and Aarhus University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
short interval intracortical inhibition (SICI) measured by threshold tracking TMS | 8 hours
  Measurement of the relative change in resting motor threshold during different interstimulus intervals and stimulus intensities
short interval intracortical inihibition (SICI) measured by conventional TMS | 8 hours
  Measurement of the size of motor evoked potentials (MEP) during different interstimulus intervals and a predetermined stimulus intensity
Concentration of GABA and glutamate | 1 hour
  Concentration of GABA and glutamate quantified as a ratio of creatine or tissue water content

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Tankisi, MD, PhD, Study Chair — Department of Clinical Neuropysiology, Aarhus University Hospital
Locations (1):
- Department of Clinical Neurophysiology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided